CLINICAL TRIAL: NCT05110703
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Assess the Safety and Effect on Quality of Life of a Prebiotic Fiber Meal Replacement Shake in Individuals With Type 2 Diabetes
Brief Title: Study to Assess Safety and Effect of a Prebiotic Fiber Meal Replacement Shake in Individuals With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uplifting Results Labs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 001-001
Record Dates: First submitted 2021-10-04; First posted 2021-11-08 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Microbiome; Fiber; Prebiotic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Nutrition Policy

STUDY DESIGN:
Intervention Model Description: This will be a 3-arm randomized, double-blinded (for the two meal replacement arms), placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary supplement: Prebiotic fiber meal replacement shake (Active Comparator): Prebiotic fiber meal replacement shake
  Interventions: Dietary Supplement: Supergut
- Dietary supplement: Placebo meal replacement shake (Placebo Comparator): Placebo meal replacement shake
  Interventions: Dietary Supplement: Placebo
- Dietary guidelines (Other): Dietary guidelines
  Interventions: Other: Dietary guidelines

INTERVENTIONS:
Dietary Supplement: Supergut — Meal replacement shake
  Arms: Dietary supplement: Prebiotic fiber meal replacement shake
Dietary Supplement: Placebo — Placebo
  Arms: Dietary supplement: Placebo meal replacement shake
Other: Dietary guidelines — Dietary guidelines
  Arms: Dietary guidelines

SUMMARY:
This study is a double-blind, randomized, trial of a commercially available meal-replacement shake versus a placebo control designed to evaluate the impact on quality of life, safety, and tolerability. It also includes a randomized, non-blinded third arm consisting of only dietary guidelines.

DETAILED DESCRIPTION:
A total of 147 participants will be recruited for the study following screening, with the expectation that approximately 131 participants will complete the trial. The 147 participants will be randomized to the three different study arms in a 2:1:1 ratio with the commercially available meal-replacement shake group being the one favored, i.e., 73 participants in that arm and 37 in the other two arms.

The trial will be mostly virtual, with in-person visits to a laboratory facility for blood draws, as well as standardized BMI calculations, waist circumference, and blood pressure readings. A technology platform will be utilized to screen, enroll and capture study data of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2D for ≥90 days
* HbA1c of 7.5 to 10.5%, inclusive
* BMI of 27 to 50 kg/m2, inclusive
* Treatment for T2D with lifestyle intervention only (for at least 90 days) or, if using antidiabetic medication(s), treated with a stable daily dose (for at least 90 days) of any of the following agents alone or in any combination: metformin (any formulation), sulfonylurea (e.g., glyburide, glipizide, glimepiride), DPP-4 inhibitor (e.g., sitagliptin, saxagliptin, linagliptin), SGLT-2 inhibitor (e.g., empagliflozin, canagliflozin, dapagliflozin, ertugliflozin), GLP-1 receptor agonists (e.g., liraglutide, semaglutide, dulaglutide)

Exclusion Criteria:

* Have type 1 diabetes or secondary forms of diabetes (e.g., secondary to cystic fibrosis)
* Have a history of severe hypoglycemia or hyperglycemia requiring hospitalization within the prior 6 months
* Have required insulin therapy for the treatment of T2D (with the exception of prior acute, temporary use during a hospitalization and/or for past treatment of gestational diabetes)
* Treatment with any glucose-lowering agent(s) other than those stated in the inclusion criteria during a period of 90 days prior to screening
* Receiving chronic oral steroid therapy (excluding those for skin, eyes, nose, or inhaled) or have received such therapy within 1 month of screening
* Female who is pregnant, breastfeeding or intends to become pregnant during the course of the study
* Participation in a clinical research trial within 30 days prior to screening
* Food allergies to ingredients in the shake including but not limited to milk protein allergy
* Ankylosing spondylitis
* Crohn's disease
* Celiac disease
* Cardiovascular (CV) conditions within 2 months prior to screening: acute myocardial infarction, cerebrovascular accident (stroke), or hospitalization due to congestive heart failure (CHF)
* Other gastrointestinal conditions which in the investigator's opinion may jeopardize the individual's safety or interfere with the ability to comply with the study.
* Gastrointestinal surgeries such as those for weight loss, large bowel resection or small bowel resection which in the investigator's opinion may jeopardize the individual's safety or interfere with the ability to comply with the study.
* Have a history of any other condition such as known drug, alcohol abuse, or psychiatric disorder which in the investigator's opinion may jeopardize the individual's safety or interfere with the ability to comply with the study.
* Any disorder, unwillingness or inability, which in the investigator's opinion, might jeopardize the individual's safety or interfere with the ability to comply with the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Examination of the effect of daily use of a prebiotic fiber meal replacement (PFMR) shake on quality of life [Time Frame: Baseline to 12 weeks] | 12 weeks
  The endpoint will be reported by the participant on a scale to measure the quality of life. Participants will complete the surveys at baseline and 12-weeks. The study uses a questionnaire including a scale from 0-5 to assess their quality of life(0=not a problem and 5=a very serious problem).

SECONDARY OUTCOMES:
To examine the effect of PFMR shakes on hunger [Time Frame: Baseline to 12 weeks] | 12 weeks
  The endpoints will be reported by the participant as follows: Hunger: surveys at baseline and 12-weeks. The study uses a questionnaire including a scale from 0-10 to assess hunger (0=starving & beyond and 10=thanksgiving full)
Changes from baseline on gastrointestinal symptoms after daily use of PFMR shakes [Time Frame: Baseline to 12 weeks] | 12 weeks
  The endpoints will be reported by the participant as follows: Gastrointestinal symptoms: surveys at baseline and 12-weeks. The study uses a questionnaire including a scale from 0-7 to assess gastrointestinal discomfort (0=no discomfort at all and 7=very severe discomfort)
Changes from baseline in fruit, vegetable, and fiber consumption. [Time Frame: Baseline to 12 weeks] | 12 weeks
  The endpoints will be reported by the participant as follows: Fruit, vegetable, and fiber consumption: surveys at baseline and 12-weeks. The study uses a questionnaire including a scale from 0-6 to assess consumption (0=no consumption; 6=daily consumption)
Changes from baseline in A1C associated with type 2 diabetes (T2D) after daily use of PFMR shakes [Time Frame: Baseline to 12 weeks] | 12 weeks
  Changes in biomarkers associated with T2D (changes in a1c) at baseline, 4-weeks, and 12-weeks.
Changes from baseline in blood pressure after daily use of PFMR shakes on blood pressure. [Time Frame: Baseline to 12 weeks] | 12 weeks
  Changes in blood pressure at baseline, 4-weeks, and 12-weeks.
Changes from baseline in body weight after daily use of PFMR shakes. [Time Frame: Baseline to 12 weeks] | 12 weeks
  Changes in body weight (in lbs) are measured at baseline, 4-weeks, and 12-weeks.
Changes from baseline on short-chain fatty acid synthesis from baseline after daily use of PFMR shakes. [Time Frame: Baseline to 12 weeks] | 12 weeks
  Changes is short chain fatty acids synthesis measured with an at-home stool kit at baseline, 4 weeks, and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Frias, MD, Principal Investigator — Uplifting Results Labs Inc.
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided